CLINICAL TRIAL: NCT02719717
Title: Prospective, Multi-Center, International Phase 2 Trial of the Use of Ultrasonic Energy for Pulmonary Artery Branch Sealing During VATS Lobectomy
Brief Title: Ultrasonic Energy for Pulmonary Artery Branch Sealing During VATS Lobectomy
Acronym: VATS PA-ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 15.302
Record Dates: First submitted 2016-01-28; First posted 2016-03-25 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
Keywords: VATS lobectomy; vascular sealing; energy; pulmonary artery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Harmonic Ace+7 (Experimental): Pulmonary artery sealing with Harmonic Ace+7 in VATS lobectomy
  Interventions: Device: Harmonic Ace+7

INTERVENTIONS:
Device: Harmonic Ace+7 — Pulmonary artery sealing with Harmonic Ace+7 in VATS lobectomy

SUMMARY:
This research program consists of a prospective, multi-institutional Phase 2 trial and an economic cost-effectiveness analysis for the use of ACE+7 in VATS lobectomy/segmentectomy compared to traditional techniques.

It will be left up to the study credentialed surgeon investigator to decide the suitability of PA branches for sealing. This will be decided intra-operatively based on anatomy, vascular dissection and length as well as patient specific factors.

DETAILED DESCRIPTION:
Currently, a minority of anatomic pulmonary resections are being performed by VATS (15%). The technical difficulty and increased actual and perceived danger of VATS lobectomy is related to PA branch manipulation, stapling and division. This is the main limitation for many thoracic surgeons regarding the adoption of VATS lobectomy into their practice. Furthermore, the majority of VATS lobectomies are being performed in high volume, academic medical centers with a resultant disparity in socioeconomic status between those that undergo VATS versus open lobectomy. If we can find a way to decrease the manipulation required by the surgeon on the PA branches, these procedures will be safer, less stressful for the surgeon and therefore more prevalent for anatomical pulmonary resections.

Energy utilization in VATS lobectomy may also be more cost effective than endostaplers. The use of a single device for lymph node dissection, hilar dissection, and PA branch sealing may allow for overall procedural cost savings. There may also be a potential benefit in decreasing overall length of hospital stay due to decrease in chest tube duration secondary to decreased post-operative pleural fluid output following VATS lobectomy when using energy as opposed to cautery for mediastinal lymph node dissection.

Objectives:

* Systematically evaluate the immediate, short- and medium-term efficacy and safety of PA sealing utilising ACE+7 in a human VATS Lobectomy/Segmentectomy.
* Understand cost issues related to use of ACE+7 in human VATS Lobectomy/Segmentectomy.

General satisfaction of the surgeon utilizing energy sealing devices compared to standard endostaplers will be assessed using a post-procedural online survey administered by the research team immediately following each procedure.

This multi-institutional, international trial will be important to decrease the bias associated with single center studies and bolster the confidence level of thoracic surgeons in the results of the trial. Study sites have been specifically chosen in the USA, Canada and Europe in order to increase the worldwide generalizability of results.

ELIGIBILITY:
Inclusion Criteria:

1. ability to consent
2. > 18 years old
3. non-hilar tumors
4. pre-operative imaging (chest CT and PET-CT
5. invasive mediastinal staging requirement will be based on current American College of Chest Physicians (ACCP) lung cancer staging criteria and will be performed by any of the following tests, in appropriate patients, alone or in combination based on study site preference in accordance with ACCP guidelines - mediastinoscopy, mediastinotomy, VATS, endobronchial ultrasound, endoscopic ultrasound.

Exclusion Criteria:

1. previous unilateral thoracic surgical procedure or trauma
2. history of mediastinal or pulmonary irradiation
3. anticoagulation with inability to stop anticoagulants prior to surgery
4. systemic vascular disease or vasculitis
5. uncorrectable coagulopathy
6. use of systemic steroids or immunosuppressive medication Pulmonary hypertension will not be an exclusion criterion as patients with pulmonary hypertension were shown to have higher bursting pressures following PA sealing in previous studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
For technical success absence of intra-operative bleeding directly related to PA branch ACE+7 sealing on vessels ≤7mm. | Immediate, intra-operative evaluation
  All procedures will be video-recorded for intra-operative assessment of vascular manipulation, vessel sealing and bleeding episodes using high definition thoracoscope video recorder.

SECONDARY OUTCOMES:
Number of intra-operative transfusions | Immediate, intra-operative
Number of post-operative transfusions | After the surgery up to 30 days
Number of conversion to open surgery | Immediate, intra-operative
Number of intra-operative mortality | Immediate, intra-operative
Length of stay (days) | After the surgery up to 30 days
Chest tube drainage per 24-hour period (mL) | From the time of surgery to chest tube removal
Number of operative take-back for bleeding, source of bleeding | During the hospitalisation (up to 30 days)

OTHER OUTCOMES:
Number of morbidity and mortality | From time of discharge to follow up 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Monteal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Liberman M, Khereba M, Goudie E, Kazakov J, Thiffault V, Lafontaine E, Ferraro P. Pilot study of pulmonary arterial branch sealing using energy devices in an ex vivo model. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3219-23. doi: 10.1016/j.jtcvs.2014.05.089. Epub 2014 Jul 19. PMID 25125207
- [Background] Goudie E, Khereba M, Tahiri M, Hegde P, Thiffault V, Hadjeres R, Berdugo J, Ferraro P, Liberman M. Pulmonary Artery Sealing With an Ultrasonic Energy Device in Video-Assisted Thoracoscopic Surgery Lobectomy: An Animal Survival Study. Ann Thorac Surg. 2016 Oct;102(4):1088-94. doi: 10.1016/j.athoracsur.2016.04.050. Epub 2016 Jun 24. PMID 27345091
- [Result] Liberman M, Khereba M, Nasir B, Goudie E, Danino A, Giot JP, Nizard N, Hadjeres R, Thiffault V, Farrenq N, Ferraro P. Pulmonary Artery Sealing Using the HARMONIC ACE+ Shears for Video-Assisted Thoracoscopic Surgery Lobectomy. Ann Thorac Surg. 2015 Sep;100(3):898-903; discussion 903-4. doi: 10.1016/j.athoracsur.2015.04.063. Epub 2015 Jul 21. PMID 26209484
- [Derived] Liberman M, Goudie E, Morse C, Hanna W, Evans N, Yasufuku K, Sampalis J; VATS PA Study Working Group. Prospective, multicenter, international phase 2 trial evaluating ultrasonic energy for pulmonary artery branch sealing in video-assisted thoracoscopic surgery lobectomy. J Thorac Cardiovasc Surg. 2020 Jan;159(1):301-311. doi: 10.1016/j.jtcvs.2019.09.061. Epub 2019 Sep 30. PMID 31679701